CLINICAL TRIAL: NCT06238453
Title: The Effect of Health Belief Model-based Education Given Through Whatsapp Application on Health Beliefs Regarding Mammography and Re-mammography
Brief Title: The Effect of Training Given by Whatsapp Application on Mamography Health Beliefs and Behaviors
Status: Not yet recruiting | Type: Observational
Sponsor: Kemal Yaran (Other)
Responsible Party: Sponsor-Investigator, Kemal Yaran, Academician (Lecturer), Muş Alparslan University
Organization: Muş Alparslan University (Other)
Other Study IDs: B.30.2.ATA.0.01.00/681
Record Dates: First submitted 2023-12-29; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Health Belief Model; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Educational content will be sent to the experimental group once a week via the WhatsApp application, and individual counseling will be provided by answering their questions at the same time. A total of 8 weeks of intervention will be implemented, training will be given with training presentations in the first 6 weeks and training videos will be sent in the last 2 weeks.
- Control group: The control group will be invited to KETEM to have a mammogram without any intervention.

SUMMARY:
It is known that the healing process of breast cancer is accelerated thanks to the early diagnosis and effective treatment. Mammography screening is an important diagnostic method in the early diagnosis of breast cancer. It is thought that the education to be given according to the Health Belief Model will make important contributions to developing a positive attitude in breast cancer screenings and regular mammography.

DETAILED DESCRIPTION:
The research will consist of women who have previously applied to Erzurum Cancer Early Diagnosis, Screening and Education Center, had mammography taken, and whose phone records are available, whose appointment has been made since December 2022, and who meet the screening selection criteria. Women who have had a mammography appointment from KETEM and have not taken it yet, request their phone information. After the women were searched one by one to identify those who fit their characteristics and volunteers, they would leave the simple random experiment control elements. During the searches, all women will be invited to KETEM to have a mammogram again. The experimental group will send educational content through the WhatsApp application once a week, and will also answer questions and provide individual counseling. A total of 8 weeks of intervention will be implemented, the first 6 weeks of training will be provided with training presentations and the last 2 weeks of training video will be sent. Feedback will be received after the training presentations are followed through the WhatsApp application where they are read. The control group will not take any action and will be invited to KETEM for mammography. Pre-test and post-analysis phone access will be collected. At the end of the training, he will have the final examinations applied after 3 months. The number of women who participated in the study will be determined by examining the KETEM records of mammography.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 40-69,
* Be woman,
* Not having been diagnosed with breast cancer,
* Not to be pregnant, lactating or puerperal,
* Absence of a mental illness
* At least 2 years have passed since the last mammogram,
* Being able to use the WhatsApp application

Exclusion Criteria:

* Having had problems with breast cancer before,
* Having a mammogram at regular intervals,
* Having had breast-conserving surgery for any purpose.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of women who have applied to Erzurum Cancer Early Diagnosis, Screening and Training Center before, had mammography and phone records, whose appointment has been made since December 2022, and who meet the sampling selection criteria.
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Pre-test evaluation | Three month
  The Health Belief Model Scale for Breast Cancer Screening and the Mammography Self-Efficacy Scale will be administered to all women in the experimental and control groups for pre-test purposes. There is no overall total score of the Health Belief Model Scale on Breast Cancer Screenings. Each sub-dimension's own total score is evaluated. The scale is a Likert type scale scored from 1 to 5. The scoring of the scale ranges from 1 point for "strongly disagree" to 5 points for "strongly agree". Increasing scores obtained from sub-dimensions indicate that the perception of that sub-dimension is high. Mammography Self-Efficacy Scale has ten items and five-point Likert type. The scale answers "strongly disagree" are evaluated as 1 point, "disagree" as 2 points, "undecided" as 3 points, "agree" as 4 points and "strongly agree" as 5 points. A higher score for each dimension indicates a higher probability of having a mammogram.
Posttest evaluation | Six month
  Training presentations will be sent to the experimental group in the first 6 weeks and training videos will be sent in the last 2 weeks. A total of 8 weeks of intervention will be implemented. Training content will be sent via WhatsApp application once a week. No intervention will be made to the control group by the researchers during this period. Those in the control group will be invited to KETEM to have a mammogram. Three months after the training is completed, the Health Belief Model Scale for Breast Cancer Screening and the Mammography Self-Efficacy Scale will be administered to both groups for posttest purposes.